CLINICAL TRIAL: NCT02818153
Title: Validation of an Allergic Rhinitis Control Test in Teenagers
Acronym: ARCTado
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 9614
Record Dates: First submitted 2016-06-27; First posted 2016-06-29 (Estimated); Last update posted 2016-06-29 (Estimated); Status verified 2016-06

CONDITIONS: Allergic Rhinitis
Keywords: Allergic rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- questionnaire for allergic rhinitis control (Experimental): Teenagers from 12 to 17 years old who complete a Self questionnaire regarding allergic rhinitis control during the consultation and after 15 days
  Interventions: Other: Self questionnaire for allergic rhinitis control

INTERVENTIONS:
Other: Self questionnaire for allergic rhinitis control

SUMMARY:
Allergic rhinitis is a common condition that affects adults as well as children and adolescents, often with impaired quality of life. Patients often report a poor level of satisfaction with the effectiveness of their treatment and are always looking for more drug combinations to improve their symptom. Several tools exist for assessing control of allergic rhinitis, but none has been validated in adolescents or in children. A study conducted in 2008, resulted in the validation of a self-administered control test of allergic rhinitsis (ARCT) in patients from 12 years of age. However, this study included only 67 adolescents aged 12 to 17 years old and lacked power.

In this new study,the investigators propose, following exactly the same procedure as the pilot study of 2008, to confirme the validation of unmodified Adult questionnaire in adolescents 12 to 17 years inclusive.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 12 to 17 years old, consulting a practitioner for an allergic rhinitis
* parents formulated their study participation agreement by signing the consent form.

Exclusion Criteria:

* Patients that are already treated for the actual episode of allergic rhinitis and are satisfied of the treatement.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 200 (Estimated)
Dates: Start 2016-06; Primary Completion 2016-09 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Score of the allergic rhinitis control self questionnaire in teenagers from 12 to 17 years old. | 15 days

CONTACTS AND LOCATIONS:
Locations (1):
- University hospital of Montpellier, Montpellier, France

IPD SHARING:
Plan to Share IPD: No